

#### STATISTICAL ANALYSIS PLAN

Study Title: An Open-label Study to Assess the Long-term Safety and

Efficacy of Tirabrutinib in Subjects with Relapsed/Refractory

**B-cell Malignancies** 

Name of Test Drug: Tirabrutinib (GS-4059)

Study Number: GS-US-401-1787

**Protocol Version (Date):** Amendment 5 (29 October 2019)

**Analysis Type:** Final Analysis

**Analysis Plan Version:** Version 3.0

**Analysis Plan Date:** 10 February 2021

Analysis Plan Authors: PPD

CONFIDENTIAL AND PROPRIETARY INFORMATION

# **TABLE OF CONTENTS**

| TAI | BLE OF | F CONTENTS | 2 |
|---|---|---|---|
| LIS | T OF A | BBREVIATIONS | 5 |
| 1. | INTR | ODUCTION | 7 |
| | 1.1. | Study Objectives | 7 |
| | 1.2. | Study Design | |
| | 1.2. | 1.2.1. Study ONO-4059POE001 (Parent Study) | |
| | | 1.2.2. Study US-US-401-1787 (Rollover Study) | |
| | 1.3. | Sample Size and Power | |
| 2. | TYPE | E OF PLANNED ANALYSIS | 9 |
| | 2.1. | Interim Analyses | 9 |
| | 2.2. | Final Analysis | |
| | 2.3. | Follow-Up Analysis | |
| 3. | GENI | ERAL CONSIDERATIONS FOR DATA ANALYSES | 10 |
| | 3.1. | Analysis Sets | 10 |
| | | 3.1.1. All Enrolled Analysis Set | |
| | | 3.1.2. Full Analysis Set. | |
| | | 3.1.3. Safety Analysis Set | |
| | | 3.1.4. Pharmacokinetic Analysis Set | |
| | 3.2. | Subject Grouping | |
| | 3.3. | Strata and Covariates | |
| | 3.4. | .4. Examination of Subject Subgroups | |
| | 3.5. | | |
| | 3.6. | Missing Data and Outliers | 12 |
| | | 3.6.1. Missing Data | |
| | | 3.6.2. Outliers | |
| | 3.7. | Data Handling Conventions and Transformations | |
| | 3.8. | Analysis Visit | |
| | | 3.8.1. Definition of Study Day | |
| | | 3.8.2. Analysis Visit Windows | |
| | | 3.8.3. Selection of Data in the Event of Multiple Records at Baseline | |
| | 3.9. | Changes From Protocol-Specified General Considerations | 14 |
| 4. | SUBJ | ECT DISPOSITION | 15 |
| | 4.1. | Subject Enrollment and Disposition | 15 |
| | 4.2. | Extent of Study Drug Exposure and Adherence | 15 |
| | | 4.2.1. Duration of Exposure to Study Drug | |
| | | 4.2.2. Adherence to Study Drug | |
| | 4.3. | Protocol Deviations | |
| | 4.4. | Assessment of COVID-19 Impact | 16 |
| | | 4.4.1. Study Drug or Study Discontinuation Due to COVID-19 | 17 |
| | | 4.4.2. Protocol Deviations Due to COVID-19 | |
| | | 4.4.3. Missed and Virtual Visits Due to COVID-19 | 17 |
| 5. | BASE | ELINE CHARACTERISTICS | 18 |
| | 5.1. | Demographics | 18 |
| | 5.2. | Other Baseline Characteristics | |
| | 5.3. | Medical History | |
| | 5.4. | Disease History | 18 |
| | 5.5. | Prior Treatments | 19 |

| 6. | EFFICACY ANALYSES | | | |
|---|---|---|---|---|
| | 6.1. | Defini | tion of Efficacy Endpoint | 20 |
| | 6.2. | | sis Methods for Efficacy Endpoints | |
| | | 6.2.1. | Overall Response Rate | 20 |
| | | 6.2.2. | Progression-Free Survival | 21 |
| | | 6.2.3. | Duration of Response | 22 |
| | | 6.2.4. | Overall Survival | 22 |
| 7. | SAFETY ANALYSES | | | |
| | 7.1. | 24 | | |
| | | 7.1.1. | Adverse Event Dictionary | |
| | | 7.1.2. | Adverse Event Severity | |
| | | 7.1.3. | Relationship of Adverse Events to Study Drug | |
| | | 7.1.4. | Serious Adverse Events | |
| | | 7.1.5. | Treatment-Emergent Adverse Events | |
| | | | 7.1.5.1. Definition of Treatment-Emergent Adverse Events | |
| | | | 7.1.5.2. Incomplete Dates | |
| | | 7.1.6. | Summaries of Adverse Events and Deaths | |
| | | | 7.1.6.1. Summaries of AE Incidence by Severity | |
| | | 7.1.7. | Treatment-Emergent Adverse Events of Interest | |
| | 7.2. | | atory Evaluations | |
| | | 7.2.1. | Summaries of Numeric Laboratory Results | |
| | | 7.2.2. | Graded Laboratory Values | |
| | | | 7.2.2.1. Treatment-Emergent Laboratory Abnormalities | |
| | | | 7.2.2.2. Treatment-Emergent Marked Laboratory Abnormalities | |
| | | | 7.2.2.3. Summaries of Laboratory Abnormalities | |
| | | 7.2.3. | Liver-related Laboratory Evaluations | |
| | | 7.2.4. | Shifts Relative to the Baseline Value | |
| | 7.3. Body Weight and Vital Signs | | | |
| | 7.4. Prior and Concomitant Medications | | | |
| | | 7.4.1. | Prior Medications | |
| | | 7.4.2. | Concomitant Medications | |
| | | 7.5. Electrocardiogram Results | | |
| | 7.6. Other Safety Measures | | | |
| | 7.7. | _ | es From Protocol-Specified Safety Analyses | |
| 8. | PHARMACOKINETIC ANALYSES | | | 33 |
| | 8.1. | Pharm | acokinetics (PK) Sample Collection | 33 |
| | 8.2. | | ical Analysis Methods | |
| | 8.2.1. Tirabrutinib Plasma Concentration | | 33 | |
| | 8.3. | | | |
| 9. | REFE | ERENCES | S | 34 |
| 10. | SOFTWARE | | | 35 |
| 11. | SAP REVISION | | | 36 |
| 12. | | | | |
| | | ndix 1. | COVID-19 SMQ with Broad Scope | 38 |
| | Appendix 2. | | Determining Missing and Virtual Visits Due to COVID-19 | |
| | | ndix 3. | Bleeding/Haemorrhage Medical Search Term | |
| | | | Hypersensitivity Medical Search Term | |
| | Appendix 5. | | Cytopenia Medical Search Term | 53 |

| Appendix 6. | Cardiac arrhythmia Medical Search Term. | 55 |
|-------------|---------------------------------------------|----|
| 1.1 | Rash Medical Search Term | |
| 11 | List of Laboratory Tests for Safety Summary | |

#### LIST OF ABBREVIATIONS

AE adverse event

ALT alanine aminotransferase
AST aspartate aminotransferase
ALP alkaline phosphatase

BLQ below the limit of quantitation

BMI body mass index CI confidence interval

CLL chronic lymphocytic leukemia

CR complete response
CRF case report form
CSR clinical study report

CTCAE Common Toxicity Criteria for Adverse Events

DMC data monitoring committee

DOR duration of response ECG Electrocardiogram

ECOG Eastern Corporation Oncology Group

ET early termination
FAS Full Analysis Set
Gilead Gilead Sciences
HLT high-level term
LTT lower-level term
LOQ limit of quantitation

MedDRA Medical Dictionary for Regulatory Activities

NE not evaluable

NHL non-Hodgkin's lymphoma NLP Natural Language Processing

ORR overall response rate
OS overall survival
PD progressive disease
PK pharmacokinetic
PR partial response

PFS progression-free survival

PT preferred term

Q1, Q3 first quartile, third quartile SAP statistical analysis plan

SD stable disease

SPD sum of the products of the greatest perpendicular diameters

StD standard deviation

| SAE | serious adverse event(s) |
|------|----------------------------------|
| SAP | statistical analysis plan |
| SOC | system organ class |
| TEAE | treatment-emergent adverse event |
| TFLs | tables, figures, and listings |
| ULN | upper limit of normal |
| WHO | World Health Organization |

#### 1. INTRODUCTION

This statistical analysis plan (SAP) describes the statistical analysis methods and data presentations to be used in tables, figures, and listings (TFLs) in the clinical study report (CSR) for study GS-US-401-1787. This SAP is based on the study protocol amendment 5 dated 29 October 2019 and the electronic case report form (eCRF). The SAP will be finalized before database finalization. Any changes made after the finalization of the SAP will be documented in the CSR.

#### 1.1. Study Objectives

The primary objective of this study is as follows:

• To determine the long-term safety and tolerability of tirabrutinib in subjects in a prior tirabrutinib study ONO-4059POE001 (parent study) and whose disease had not progressed on the parent study.

The secondary objective of this study is as follows:

• To determine the long term efficacy of tirabrutinib

### 1.2. Study Design

The analysis of this rollover study GS-US-401-1787 will integrate the data from the parent study. Thus, the study design of the parent study is also described in Section 1.2.1, followed by the rollover study design in Section 1.2.2.

### 1.2.1. Study ONO-4059POE001 (Parent Study)

This is an open-label Phase 1 multi-center study with a non-randomized, adaptive dose-escalating design, to investigate the safety and tolerability of tirabrutinib administered as monotherapy to subjects with relapsed/refractory NHL and CLL. Subjects with no therapy of higher priority available and for whom treatment with a BTK inhibitor is deemed appropriate will be eligible.

Tirabrutinib was administered orally at the assigned dose levels for up to 6 cycles of treatment. Each treatment cycle consists of 28 days of continuous dosing. Continuation of treatment beyond 6 cycles is possible for subjects deriving clinical benefit from the treatment. Intra-patient dose escalation or dose de-escalation after completion of the initial 6 month treatment period is allowed to provide patients with an opportunity to maximize upon their already established clinical response. Patients may receive continuous treatment until disease progression as assessed by the investigator or until experiencing an intolerable AE leading to discontinuation of drug.

CT with contrast or MRI assessment at screening served as the baseline of efficacy evaluation. The response was assessed every 3 months during the first year of treatment and then every 6 months thereafter using the appropriate response criteria for CLL and NHL.

Study ONO-4059POE001 has completed and all subjects are now off study or have rolled over to study GS-US-401-1787. The full CSR of study ONO-4059POE001 has been completed. Adverse events and laboratory abnormalities were graded using the Common Terminology for Adverse Events (CTCAE), Version 4.0, adverse events preferred terms were coded using MedDRA 18.1, and concomitant medications were coded using WHODRUG Q2-2015.

### **1.2.2.** Study US-US-401-1787 (Rollover Study)

This study is an open-label rollover study for subjects who have tolerated and achieved stable disease or responded to tirabrutinib treatment while enrolled in the parent study ONO-4059POE001.

Subjects who meet eligibility criteria will continue to receive tirabrutinib. Each cycle will consist of 28 days of therapy. If there is no evidence of disease progression by clinical assessment or by CT (or MRI), a subject may continue receiving tirabrutinib until disease progression (clinical or radiographic) for a maximum duration of 5 years from the start of this rollover study GS-US-401-1787. After discontinuation of treatment, subjects will be followed for safety for 30 days.

CT with contrast or MRI will be obtained to document disease, in accordance with the NHL and CLL response assessment guidelines. If not performed in the previous 90 days prior to Cycle 1 Day 1 on study GS-US-401-1787, CT scan with contrast or MRI will be performed between C1D1 and C1D28, and at approximately week 12 and then every 24 weeks. Bone marrow examination (core biopsy and/or aspirate as per local standard of care) will be performed for follow-up only (for both NHL and CLL subjects) if previously positive and/or to confirm CR, if physical examination and CT-scans demonstrate a CR.

#### 1.3. Sample Size and Power

The number of subjects enrolled will be determined by the number of subjects who complete a prior tirabrutinib study who are still alive without disease progression, wish to continue therapy with tirabrutinib, and meet the study entry criteria.

# 2. TYPE OF PLANNED ANALYSIS

# 2.1. Interim Analyses

No formal interim analysis is planned.

This study does not have a data monitoring committee (DMC). Therefore, no analyses will be conducted for the DMC.

# 2.2. Final Analysis

After all subjects have completed/discontinued the study, outstanding data queries have been resolved or adjudicated as unresolvable, and the data have been cleaned and finalized, the final analysis of the data will be performed.

# 2.3. Follow-Up Analysis

No follow-up analysis is planned.

#### 3. GENERAL CONSIDERATIONS FOR DATA ANALYSES

Analysis results will be presented using descriptive statistics. For categorical variables, the number, percentage, and 95% confidence intervals (CIs) on the percentage of subjects in each category will be presented; for continuous variables, the number of subjects (n), mean, standard deviation (StD), 95% CIs on the mean, median, first quartile (Q1), third quartile (Q3), minimum, and maximum will be presented.

By-subject listings will be presented for all subjects in the All Enrolled Analysis Set and sorted by subject ID number, visit date, and time (if applicable). Data collected on log forms, such as adverse events (AEs), will be presented in chronological order within subject. Age, sex at birth, race, and ethnicity for each subject will be presented in the listings, as space permits.

### 3.1. Analysis Sets

Analysis sets define the subjects to be included in an analysis. Analysis sets and their definitions are provided in this section. The analysis set will be identified and included as a subtitle of each table, figure, and listing.

For each analysis set, the number and percentage of subjects will be summarized.

A listing of reasons for exclusion from analysis sets will be provided by subject.

### 3.1.1. All Enrolled Analysis Set

The All Enrolled Analysis Set consists of all subjects who were enrolled in the GS-US-401-1787 study. This analysis set will be used for the listings.

#### 3.1.2. Full Analysis Set

The Full Analysis Set consists of all enrolled subjects who took at least 1 dose of study drug in the GS-US-401-1787 study. This analysis set will be used for the efficacy endpoints.

#### 3.1.3. Safety Analysis Set

The Safety Analysis Set includes all subjects who took at least 1 dose of study drug in the GS-US-401-1787 study. This is the primary analysis set for safety analyses.

#### 3.1.4. Pharmacokinetic Analysis Set

The Pharmacokinetic Analysis Set consists of all subjects who enrolled in the GS-US-401-1787 study and have at least 1 evaluable PK sample.

# 3.2. Subject Grouping

For analyses based on the All Enrolled Analysis Set and Full Analysis Set, subjects will be grouped according to the treatment to which they were initially assigned at the entry of GS-US-401-1787. For analyses based on the Safety Analysis Set, subjects will be grouped according to the actual treatment with the longest exposure duration in parent and rollover study.

For the PK Analysis Set, subjects will be grouped according to the actual treatment they received prior to the PK sampling time.

All analyses will be performed for CLL and NHL subjects separately, unless otherwise specified.

The applicable dose levels of tirabrutinib are:

| Dose Levels for CLL | Dose Levels for NHL |
|---------------------|---------------------|
| 20mg QD | 20mg QD |
| 40mg QD | 40mg QD |
| 80mg QD | 80mg QD |
| 160mg QD | 160mg QD |
| 320 mg QD | 320 mg QD |
| 400 mg QD | 400 mg QD |
| 500 mg QD | 480 mg QD |
| 600 mg QD | 600 mg QD |
| 300mg BID | 240mg BID |

Summary of efficacy will be presented by integrating the parent study data and rollover study data, using only subjects who rolled over to GS-US-401-1787.

Summary of safety will be presented using only subjects who rolled over to GS-US-401-1787:

- All safety summaries will be provided combining data from both parent study (ONO-4059POE001) and rollover study (GS-US-401-1787).
- Selected safety summaries will also be provided only using data from rollover study GS-US-401-1787.

#### 3.3. Strata and Covariates

This study does not use a stratified randomization schedule in enrolling subjects. No covariates will be included in efficacy and safety analyses.

# 3.4. Examination of Subject Subgroups

Due to the limited sample size at each dose level, no subgroup analysis will be performed.

#### 3.5. Multiple Comparisons

Adjustments for multiplicity will not be made, because no formal statistical testing will be performed in this study.

### 3.6. Missing Data and Outliers

### 3.6.1. Missing Data

In general, missing data will not be imputed unless methods for handling missing data are specified. Exceptions are presented in this document.

For missing last dosing date of study drug, imputation rules are described in Section 4.2, for death in Section 6.2.4, for new anticancer therapy in Section 6.2.2, for AE onset is described in Section 7.1.5.2.

#### **3.6.2. Outliers**

Unless otherwise specified, outliers will not be excluded from the analysis in general.

## 3.7. Data Handling Conventions and Transformations

In general, age (in years) on the date of the first dose of study drug in the parent study will be used for analyses and presentation in listings. If only birth year is collected on the CRF, "01 July" will be used for the unknown birth day and month for the purpose of age calculation. If only birth year and month are collected, "01" will be used for the unknown birth day.

Non-PK Data that are continuous in nature but are less than the lower limit of quantitation (LOQ) or above the upper LOQ will be imputed as follows:

- A value that is 1 unit less than the LOQ will be used for calculation of descriptive statistics if the datum is reported in the form of "< x" (where x is considered the LOQ). For example, if the values are reported as < 50 and < 5.0, values of 49 and 4.9, respectively, will be used for calculation of summary statistics. An exception to this rule is any value reported as < 1 or <0.1, etc. For values reported as < 1 or < 0.1, a value of 0.9 or 0.09, respectively, will be used for calculation of summary statistics.
- A value that is 1 unit above the LOQ will be used for calculation of descriptive statistics if the datum is reported in the form of "> x" (where x is considered the LOQ). Values with decimal points will follow the same logic as above.
- The LOQ will be used for calculation of descriptive statistics if the datum is reported in the form of " $\leq$  x" or " $\geq$  x" (where x is considered the LOQ).

If methods based on the assumption that the data are normally distributed are not adequate, analyses may be performed on transformed data or nonparametric analysis methods may be used, as appropriate.

Natural logarithm transformation will be used for plasma/blood concentrations and analysis of PK parameters. Plasma concentration values that are below the limit of quantitation (BLQ) will be presented as "BLQ" in the concentration data listing. Values that are BLQ will be treated as 0 at predose time points, and one-half the value of the LOQ at postbaseline time points, where LOQ is corrected for the dilution factor (ie, reported LOQ/dilution factor) for determination of summary and order statistics.

The following conventions will be used for the presentation of summary and order statistics:

- If at least 1 subject has a concentration value of BLQ for the time point, the minimum value will be displayed as "BLQ."
- If more than 25% of the subjects have a concentration data value of BLQ for a given time point, the minimum and Q1 values will be displayed as "BLQ."
- If more than 50% of the subjects have a concentration data value of BLQ for a given time point, the minimum, Q1, and median values will be displayed as "BLQ."
- If more than 75% of the subjects have a concentration data value of BLQ for a given time point, the minimum, Q1, median, and Q3 values will be displayed as "BLQ."
- If all subjects have concentration data values of BLQ for a given time point, all order statistics (minimum, Q1, median, Q3, and maximum) will be displayed as "BLQ."

#### 3.8. Analysis Visit

#### 3.8.1. Definition of Study Day

Study day will be calculated from the first dosing date of study drug in parent study ONO-4059POE001 and derived as follows:

- For postdose study days: Assessment Date First Dosing Date + 1
- For days prior to the first dose: Assessment Date First Dosing Date

Therefore, study day 1 is the day of first dose of study drug administration in the parent study.

#### 3.8.2. Analysis Visit Windows

Baseline is defined as the last nonmissing value on or prior to first dosing date of study drug, unless specified differently.

For postbaseline, nominal visit as recorded on the CRF will be used when data are summarized by visit, if any. Any data relating to unscheduled visits will not be assigned to a particular visit or time point. However, the following exceptions will be made:

- An unscheduled visit prior to the first dosing of study drug may be included in the calculation of the baseline value, if applicable.
- Unscheduled visits after the first dose of study drug will be included in order to determine the maximum post-baseline toxicity grade.

# 3.8.3. Selection of Data in the Event of Multiple Records at Baseline

For baseline, the last nonmissing value on or prior to first dosing date of study drug will be selected, unless specified differently. If there are multiple records with the same time or no time recorded on the same day, the baseline value will be the average of the measurements for continuous data, or the measurement with the lowest severity (eg, normal will be selected over abnormal for safety electrocardiogram [ECG] findings) for categorical data.

### 3.9. Changes From Protocol-Specified General Considerations

In protocol, the Full Analysis Set is defined as all subjects who enrolled and treated in the parent study, and will be used for the safety and efficacy endpoints analysis. Given the study objective is to determine the long-term safety and efficacy in subjects who were in the parent study and whose disease had not progressed on the parent study (a.k.a. the rollover patient), analysis only include these rollover patient is better aligned with the study objective. Thus, in this SAP, the efficacy and safety analysis will only include subjects who enrolled in the GS-US-401-1787 study as specified in Section 3.1 and Section 3.2.

#### 4. SUBJECT DISPOSITION

### 4.1. Subject Enrollment and Disposition

A summary of subject enrollment will be provided by disease type (CLL, NHL) and dose level for each country, investigator, and overall as specified in Section 3.2 using All Enrolled Analysis Set. The summary will present the number and percentage of subjects enrolled. For each column, the denominator for the percentage calculation will be the total number of subjects analyzed for that column.

This summary will present the number of subjects screened, the number of subjects who met all eligibility criteria but were not enrolled with reasons subjects not enrolled, the number of subjects enrolled, and the number of subjects in each of the categories listed below:

- Enrolled in Study GS-US-401-1787
- Treated in Study GS-US-401-1787
- Completed study drug per protocol specified duration
- Discontinued study drug in GS-US-401-1787 with reason
- Discontinued Study GS-US-401-1787 with reasons

For the status of study drug and study completion and reasons for discontinuation, the number and percentage of subjects in each category will be provided. The denominator for the percentage calculation will be the total number of subjects in the All Enrolled Analysis Set corresponding to that column. In addition, a flowchart will be provided to depict the disposition.

A by-subject listing will be provided by subject identification (ID) number in ascending order to support the above summary table.

#### 4.2. Extent of Study Drug Exposure and Adherence

Extent of exposure to study drug will be examined by assessing the total duration of exposure to study drug and the level of adherence relative to the study drug regimen specified in the protocol.

#### 4.2.1. Duration of Exposure to Study Drug

Total duration of exposure to study drug will be defined as last dosing date minus first dosing date plus 1, regardless of any temporary interruptions in study drug administration, and will be expressed in weeks and cycles using up to 1 decimal place (eg, 4.5 weeks). If the last study drug dosing date is missing, the following imputation rule will be applied:

• If the study drug is permanently withdrawn, the latest date among the study drug end date, clinical visit date, laboratory sample collection date, and vital signs assessment date will be used.

The total duration of exposure to study drug and the total number of cycles a subject was exposed to study drug, and number and percentage of subjects who have dose reduction or interruptions will be summarized using descriptive statistics. The number (ie, cumulative counts) and percentage of subjects exposed to study drug will be summarized by cycle, where each cycle consists of 28 days of therapy. Summaries will be provided by dose level for the Safety Analysis Set.

No formal statistical testing is planned.

### 4.2.2. Adherence to Study Drug

ONO-4059POE001 collected number of doses dispensed but didn't collect dose strength of the drug kit. GS-US-401-1787 collected number of tablets/capsules dispensed but subjects may receive different strength of tablets/capsules throughout the study. Due to the inconsistent way of drug dispensation data collection in the two studies, it's not feasible to track total number of doses or total amount drug administered. Thus, drug adherence analysis will not be performed.

A by-subject listing of study drug administration and drug accountability will be provided by subject ID number (in ascending order), and visit (in chronological order).

A by-subject listing of study drug administration for subjects with dose modifications at any time will also be provided.

#### 4.3. Protocol Deviations

Subjects who did not meet the eligibility criteria for study entry, but enrolled in the study will be summarized regardless of whether they were exempted by the sponsor or not. The summary will present the number and percentage of subjects who did not meet at least 1 eligibility criterion and the number of subjects who did not meet specific criteria by disease and dose level based on the All Enrolled Analysis Set. A by-subject listing will be provided for those subjects who did not meet at least 1 eligibility (inclusion or exclusion) criterion. The listing will present the eligibility criterion (or criteria if more than 1 deviation) that subjects did not meet and related comments, if collected.

Protocol deviations occurring after subjects entered the study are documented during routine monitoring. The number and percentage of subjects with important protocol deviations by deviation reason (eg, nonadherence to study drug, violation of select inclusion/exclusion criteria) will be summarized by disease type and dose level for the All Enrolled Analysis Set. A by-subject listing will be provided for those subjects with important protocol deviation and will be sorted by subject ID number (in ascending order), and visit (in chronological order).

#### 4.4. Assessment of COVID-19 Impact

This study was ongoing during the novel coronavirus (2019 nCOV [COVID-19]) pandemic, and the COVID-19 pandemic has caused a disruption in the regular visit schedules for this study. Some subjects were unable to attend onsite visits due to shelter in place guidelines, site closures,

or other reasons. This section provides how to handle special situations due to COVID-19 in the analysis.

Adverse events (AEs) due to COVID-19 will be included in AE analyses if applicable. A bysubject listing of Adverse Events due to COVID-19 may be provided. The COVID-19 Standardized MedDRA Queries (SMQ) with Broad Scope in Appendix 1 will be implemented.

### 4.4.1. Study Drug or Study Discontinuation Due to COVID-19

A by-subject listing of reasons for premature study drug or study discontinuation due to COVID-19 will be created.

#### 4.4.2. Protocol Deviations Due to COVID-19

A by-subject listing will be provided for subjects with important protocol deviation related to COVID-19. A separate listing will be provided for subjects with non-important protocol deviation related to COVID-19.

#### 4.4.3. Missed and Virtual Visits Due to COVID-19

A by-subject listing of subjects with missed or virtual visits due to COVID-19 will be provided by subject ID number in ascending order .

Information regarding virtual or missed visits due to COVID-19 was collected as free text in the CRF comment fields. The determination of missing or virtual visits due to COVID-19 was done using Natural Language Processing (NLP) to search the CRF comment fields. A detailed explanation of the algorithm is given in Appendix 2.

#### 5. BASELINE CHARACTERISTICS

# 5.1. Demographics

Subject demographic variables (ie, age, sex, race, and ethnicity) were collected in the parent study, and will be summarized by disease type and dose level using descriptive statistics for age, and using number and percentage of subjects for sex, race, and ethnicity. The summary of demographic data will be provided for the FAS.

A by-subject demographic listing, including the informed consent date, will be provided and sorted by subject ID number in ascending order.

#### **5.2.** Other Baseline Characteristics

Other baseline characteristics include body weight (in kg), height (in cm), body mass index (BMI; in kg/m²), and ECOG Performance Status. These baseline characteristics were collected in the parent study, and will be summarized by disease type and dose level using descriptive statistics for continuous variables and using number and percentage of subjects for categorical variables. The summary of baseline characteristics will be provided for the FAS. No formal statistical testing is planned.

A by-subject listing of other baseline characteristics will be provided and sorted by subject ID number in ascending order.

#### 5.3. Medical History

Medical history will be based on data collected in the parent study, and ongoing AE from the parent study collected as general medical history in the rollover study.

Medical history data in the rollover study will not be coded. All medical history data including parent and rollover study will be listed only.

#### 5.4. Disease History

The disease history was collected in the parent study. A summary of disease-specific medical history will be provided for the Full Analysis Set.

Time since initial diagnosis (years) will be calculated as (first dosing date of study drug – date of initial diagnosis + 1) / 365.25. Time since initial diagnosis will be summarized using descriptive statistics for a continuous variable.

Disease stage at screening will be summarized using number and percentage of subjects. History of the disease staging or prognostic characterization including FLIPI (follicular lymphoma international prognostic index), IPI (international prognostic index), or MIPI (Mantle cell lymphoma International prognostic index) for NHL subjects and Binet/Rai staging for CLL subjects, will be summarized.

NHL disease subtypes (Diffuse Large B Cell Lymphoma [DLBCL], Mantle Cell Lymphoma [MCL], Follicular Lymphoma [FL], Small Lymphocytic Lymphoma [SLL], Waldenstrom's macroglobulinemia [WM], and Other) as well as DLBCL subtypes will be summarized.

The DLBCL category may be further broken down to

- DLBCL (ABC)
- DLBCL (GCB)
- DLBCL (other non-specified)

For CLL subjects, disease will be classified according to results for CLL prognostic markers as:

- 11q deletion (yes/no)
- 17p deletion (yes/no)
- TP53 mutation (yes/no)
- IgVh mutation (yes/no)

For both NHL and CLL, disease will also be classified based on response to last treatment as:

- Refractory
- Relapsed

A listing of disease-specific history will be provided.

#### 5.5. Prior Treatments

Prior treatments including prior systemic therapy, radio therapies, transplants and surgeries are collected in the parent study. The number of prior treatments a subject used in each of these categories will be summarized by disease type and dose level using the FAS.

A listing will be provided for each category of the prior treatments.

#### 6. EFFICACY ANALYSES

## 6.1. Definition of Efficacy Endpoint

Subjects' efficacy data will be integrated with the parent study as specified in Section 3.2. The efficacy analysis will be based on FAS defined in Section 3.1.2.

The efficacy endpoints are:

- Overall response rate (ORR): defined as the proportion of subjects who achieve partial response (PR) or complete response (CR) in either the parent or roll-over study
- Progression free survival (PFS): defined as the interval from date of the first dose of tirabrutinib on the parent study to the earlier of the first documentation of definitive disease progression as assessed by the investigator, or death from any cause
- Duration of response (DOR): defined as the interval from first documentation of CR or PR to the earlier of the first documentation of definitive disease progression as assessed by the investigator, or death from any cause in subjects who achieve a response.
- Overall Survival (OS): defined as the interval from date of the first dose of tirabrutinib on the parent study until death from any cause

The response or definitive disease progression for ORR, PFS, and DOR are based on the Modified IWCLL Criteria {Hallek 2008} for CLL subjects and standardized response criteria for malignant lymphoma for NHL subjects {Cheson 2007, Owen 2013}.

#### 6.2. Analysis Methods for Efficacy Endpoints

### **6.2.1.** Overall Response Rate

Best overall response (BOR) is defined as the best response recorded after first dose and prior to the time of initiation of anti-cancer therapy other than the study treatment. BOR could be assessed as CR, PR, Stable Disease (SD), or Progressive Disease (PD). In addition, a response category of Not Evaluable (NE) is provided for situation in which there is inadequate information to otherwise categorize response status.

Based on the investigator assessments, the following will be performed for the FAS by disease type and dose level:

- BOR will be summarized using the number and the percentage of subjects in each category.
- ORR will be presented with corresponding 2-sided 95% exact confidence intervals (CIs) based on Clopper-Pearson method. Subjects who do not have sufficient baseline or on-study tumor assessments to characterize response will be counted as non-responders and included in the denominator in calculate of response rates.

A by-subject listing of response will be provided by subject ID and by visit in ascending order. A by-subject listing of bone marrow results for those with CR will be provided by subject ID and by visit in ascending order.

### **6.2.2.** Progression-Free Survival

The date of definitive progression will be the time point at which progression is first identified by relevant radiographic, imaging, or clinical data. Subjects without progression or death will be censored at the last adequate post-baseline tumor assessment time. If subjects received the anticancer therapy or have  $\geq 2$  consecutive missing post-baseline tumor assessments immediately before documented progression or death, they will be censored at the last adequate post-baseline tumor assessment time before starting anti-cancer therapy or before  $\geq 2$  consecutive missing assessments, whichever is earlier. If subjects don't have an adequate baseline tumor assessment or any adequate post-baseline tumor assessments, they will be censored on the date of Study Day 1 unless they died before or on the 2nd scheduled post-baseline tumor assessment without receiving anti-cancer therapy.

PFS in months = (date of event/censoring - date of first dose + 1) / 30.4375.

When imaging examinations for one visit are conducted on various dates, the following rules apply for the calculation of the assessment date:

- The response date will be the last date associated with that particular imaging time point.
- The progression date will be the first date associated with that particular imaging time point.

When the date of initiation of anticancer therapy other than the study treatment is incomplete or missing, the following algorithm will be followed:

- If the day is missing but the month and year are available, then the imputed day will be the first day of the month.
- If day and month are missing but year is available, then the imputed day and month will be 01Jan or the last day of the month for the last adequate disease assessment if they have the same year, whichever is later.

In case that PFS event is a death with incomplete date, the imputation algorithm is as specified in section 6.2.4.

The analysis of PFS will be performed using the Kaplan-Meier method for FAS. Medians, Q1, Q3, the proportion of subjects who are progression-free at 6, 12, 18, 24, 30, 36, 42, 48, and 60 months from Study Day 1 will be provided along with corresponding 95% CIs. Kaplan-Meier curves will be provided.

The follow-up time for PFS, defined as the interval from the first dosing date of study drug to the loss to PFS follow-up, will be summarized by treatment groups using statistics such as median,

Q1, Q3 with corresponding 95% CIs estimated with the reverse K-M method. The reverse K-M model switches the event/censoring indicators of subjects in the original PFS analysis with Kaplan-Meier method. It considers subjects lost to PFS follow-up as achieving the full follow-up, and the full follow-up time of those subjects who had disease progression or died could not be observed as it is "censored" by the event.

A listing will be provided for the information of subject PFS, date of progression or censor, and reason.

A listing will be provided for the information of post-treatment anticancer therapy.

### **6.2.3. Duration of Response**

DOR will be evaluated using investigator assessments based on subset of FAS subjects who achieve a CR or PR and maintain the response. DOR will be summarized using Kaplan-Meier methods (median, Q1, Q3, and corresponding 95% CI). The same censoring rules as for PFS will be applied to DOR.

DOR in months = (date of event/censoring - date of first response [CR or PR] + 1) / 30.4375.

A by-subject listing of DOR will be provided by subject ID number in ascending order.

#### 6.2.4. Overall Survival

Subjects who are lost to follow-up or survived until the end of study will be censored at the last date that they were known to be alive.

Every attempt will be made to ensure that complete death dates are recorded. In those rare instances where complete death dates are not recorded, the following algorithm will be used:

- If day is missing but the month and year are available, then the imputed date will be the 1<sup>st</sup> day of the month or the last known alive date + 1, whichever is later.
- If day and month are missing but year is available, then the imputed date and month will be 01Jan or the last known alive date + 1, whichever is later.

If the last known alive date is not complete, the following algorithm will be used:

- If day is missing but the month and year are available, then the imputed date will be the 1st day of the month.
- If day and month are missing but year is available, then the imputed date and month will be 01Jan

The analysis of OS will be performed using the Kaplan-Meier method for FAS. Medians, Q1, Q3, the proportion of subjects who are alive at 6, 12, 18, 24, 30, 36, 42, 48, and 60 months from Study Day 1 will be provided along with corresponding 95% CIs. Kaplan-Meier curves will be provided. A listing will be provided for the information of subject OS, date of death or censor, and reason.

The follow-up time for OS, defined as the interval from the first dosing date of study drug to the loss to follow-up, will be summarized by treatment groups using statistics such as median, Q1, Q3 with corresponding 95% CIs estimated with the reverse Kaplan-Meier (K-M) method. The reverse K-M model switches the event/censoring indicators of subjects in the original OS analysis with Kaplan-Meier method. It considers subjects lost to follow-up as achieving the full follow-up, and the full follow-up time of those subjects who died could not be observed as it is "censored" by death.

#### 7. SAFETY ANALYSES

As specified in Section 3.2, subjects' safety data of GS-US-401-1787 will be integrated with the parent study for all safety analysis. Some selected safety summaries will also be provided only using data from rollover study GS-US-401-1787.

#### 7.1. Adverse Events and Deaths

#### 7.1.1. Adverse Event Dictionary

Clinical and laboratory adverse events (AEs) for the rollover study GS-US-401-1787 will be coded using the current version of MedDRA. The coding of clinical and laboratory adverse events for the completed parent study ONO-4059POE001 will be upversioned to the current version of MedDRA, and integrated with GS-US-401-1787 for analysis. System organ class (SOC), high-level group term (HLGT), high-level term (HLT), preferred term (PT), and lower-level term (LLT) will be provided in the AE dataset.

#### 7.1.2. Adverse Event Severity

Adverse events are graded by the investigator as Grade 1, 2, 3, 4, or 5 according to CTCAE Version 4.03 in 401-1787, and CTCAE Version 4.0 in ONO-4059POE001. The severity grade of events for which the investigator did not record severity will be categorized as "missing" for tabular summaries and data listings. The missing category will be listed last in summary presentation.

#### 7.1.3. Relationship of Adverse Events to Study Drug

Related AEs are those for which the investigator selected "Related" on the AE case report form (CRF) to the question of "Related to Study Treatment." Relatedness will always default to the investigator's choice, not that of the medical monitor. Events for which the investigator did not record relationship to study drug will be considered related to study drug for summary purposes. However, by-subject data listings will show the relationship as missing.

#### 7.1.4. Serious Adverse Events

Serious adverse events (SAEs) will be identified and captured as SAEs if AEs met the definitions of SAE that were specified in the study protocol. Serious adverse events captured and stored in the clinical database will be reconciled with the SAE database from the Gilead Pharmacovigilance and Epidemiology Department before data finalization.

# 7.1.5. Treatment-Emergent Adverse Events

### 7.1.5.1. Definition of Treatment-Emergent Adverse Events

Treatment-emergent adverse events (TEAEs) are defined as one or both of the following:

- Any AEs with an onset date on or after the study drug start date of parent study and no later than 30 days after permanent discontinuation of study drug
- Any AEs leading to premature discontinuation of study drug.

#### 7.1.5.2. Incomplete Dates

In case when the AE onset date is incomplete and needs to be imputed, the following algorithm will be followed:

- If the day is missing but the month and year are available, then the imputed day will be the first day of the month or the first dosing date if they have the same month and year, whichever is later.
- If the day and month are missing but year is available, then the imputed day and month will be 01Jan or the first dosing date if they have the same year, whichever is later.

An AE with completely missing onset and stop dates, or with the onset date missing and a stop date later than the first dosing date of study drug, will be considered to be treatment emergent. In addition, an AE with the onset date missing and incomplete stop date with the same or later month and year (or year alone if month is not recorded) as the first dosing date of study drug will be considered treatment emergent.

#### 7.1.6. Summaries of Adverse Events and Deaths

Treatment-emergent AEs will be summarized based on the Safety Analysis Set.

#### 7.1.6.1. Summaries of AE Incidence by Severity

The number and percentage of subjects who experienced at least 1 TEAE will be provided and summarized by SOC, PT, and dose level. For other AEs described below, summaries will be provided by SOC, PT, maximum severity and dose level:

- TEAEs
- TEAEs of Grade 3 or higher
- TE Treatment-related TEAEs
- TE Treatment-related TEAEs of Grade 3 or higher

- TE SAEs
- TE treatment-related SAEs
- TEAEs leading to dose modification of study drug
- TEAEs leading to temporary interruption of study drug
- TEAEs leading to discontinuation of study drug
- TEAEs leading to discontinuation of study
- TEAEs leading to death

A brief, high-level summary of AEs described above will be provided by dose level and by the number and percentage of subjects who experienced the above AEs. In addition, all death will also be included in this high-level summary.

In addition, TEAE by PT only will also be summarized.

In addition to the above summary tables, the following AE tables will also be provided using different grouping rule or data scope:

| Data Scope | Grouping Rule | AE Summaries |
|---|---|---|
| Integrate data from both<br>ONO-4059POE001 and GS-US-401-<br>1787 | Combine all subjects regardless of disease type or dose level | Brief high-level summary of AE<br>TEAE, TEAEs of Grade 3 or higher, SAE,<br>TEAE leading to death by SOC, PT, and<br>Severity |
| Only data from GS-US-401-1787 | Separate table by NHL and CLL Combine all subjects regardless of disease type or dose level | Brief high-level summary of AE<br>TEAE, TEAEs of Grade 3 or higher, SAE,<br>TEAE leading to death by SOC, PT, and<br>Severity |

Multiple events will be counted only once per subject in each summary. Adverse events will be summarized and listed first in alphabetic order of SOC, and then by PT in descending order of total frequency within each SOC. For summaries by severity grade, the most severe grade will be used for those AEs that occurred more than once in an individual subject during the study.

In addition, data listings will be provided for the following:

- All AEs
- All AEs of Grade 3 or higher
- SAEs

- AEs leading to death
- Deaths
- AEs leading to discontinuation of study drug
- AEs leading to dose modifications or temporary interruption of study drug
- AEs leading to discontinuation of study

#### 7.1.7. Treatment-Emergent Adverse Events of Interest

The treatment-emergent AEs of interest (AEI) include:

| AEI | Grouped Terms |
|---|---|
| Hemorrhage/Bleeding | MST-CT Bleeding/Haemorrhage (Appendix 3) |
| Infections | SOC: Infections and infestations |
| Hypersensitivity | MST-CT Hypersensitivity (Appendix 4) |
| Cytopenia | MST: Anemia-related events, leukopenias, neutropenia, thrombocytopenias (Appendix 5) |
| Cardiac Arrhythmias | MST-CT Cardiac arrhythmia and bradycardia_narrow (Appendix 6) |
| Diarrhoea | PT: Diarrhoea |
| Rash | MST-CT Rash - specific to ONC (Appendix 7) |

The following summaries will be provided for AEIs by SOC, PT, and maximum severity:

- TEAE
- TEAEs leading to dose modifications or temporary interruption of study drug
- TEAEs leading to discontinuation of study drug

A data listing of AEIs will be provided by alphabetic ascending order of AEI name, then by subject ID.

### 7.2. Laboratory Evaluations

Laboratory data collected during the study will be analyzed and summarized using both quantitative and qualitative methods. Summaries of laboratory parameters listed in Appendix 8 will be provided for the Safety Analysis Set and will include data collected up to the last dose of study drug plus 30 days for subjects who have permanently discontinued study drug. The analysis will be based on values reported in conventional units. When values are below the LOQ, they will be listed as such, and the closest imputed value will be used for the purpose of calculating summary statistics as specified in Section 3.7.

A by-subject listing for laboratory test results will be provided by subject ID number and time point in chronological order for hematology, serum chemistry, and urinalysis separately. Values falling outside of the relevant reference range and/or having a severity grade of 1 or higher on the CTCAE severity grade will be flagged in the data listings, as appropriate.

No formal statistical testing is planned.

## 7.2.1. Summaries of Numeric Laboratory Results

Descriptive statistics of selected laboratory results will be provided by treatment group as follows:

- Baseline values
- Postbaseline maximum
- Postbaseline minimum
- Change from baseline to postbaseline maximum
- Change from baseline to postbaseline minimun

A baseline laboratory value will be defined as the last measurement obtained on or prior to the date/time of first dose of study drug in parent study. Change from baseline to a postbaseline visit will be defined as the visit value minus the baseline value. Laboratory test results collected at unscheduled visits will be included for the baseline and postbaseline maximum and minimum value selection. The mean, median, Q1, Q3, minimum, and maximum values will be displayed to the reported number of digits; StD values will be displayed to the reported number of digits plus 1.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3.

# 7.2.2. Graded Laboratory Values

CTCAE Version 4.03 will be used for assigning toxicity grades (0 to 4) to laboratory results for analysis. Grade 0 includes all values that do not meet the criteria for an abnormality of at least Grade 1. For laboratory tests with criteria for both increased and decreased levels, analyses for each direction (ie, increased, decreased) will be presented separately.

#### 7.2.2.1. Treatment-Emergent Laboratory Abnormalities

Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study drug plus 30 days for subjects who permanently discontinued study drug. If the relevant baseline laboratory value is missing, any abnormality of at least Grade 1 observed within the time frame specified above will be considered treatment emergent. Local labs will be graded based on the central lab normal ranges with in-house macro. In the event that both central and local lab results are collected in the clinical database, the worst toxicity grade will be used for the summary of lab toxicities. All central and local laboratory values will be listed.

# 7.2.2.2. Treatment-Emergent Marked Laboratory Abnormalities

Treatment-emergent marked laboratory abnormalities are defined as values that increase from baseline by at least 3 toxicity grades at any postbaseline time point, up to and including the date of the last dose of study drug plus 30. If the relevant baseline laboratory value is missing, any Grade 3 or 4 values observed within the timeframe specified above will be considered treatment-emergent marked abnormalities.

### 7.2.2.3. Summaries of Laboratory Abnormalities

The following summaries (number and percentage of subjects) for treatment-emergent laboratory abnormalities will be provided by lab test and treatment group; subjects will be categorized according to the most severe postbaseline abnormality grade for a given lab test:

- Graded laboratory abnormalities
- Grade 3 or 4 laboratory abnormalities
- Marked laboratory abnormalities

For all summaries of laboratory abnormalities, the denominator is the number of subjects with nonmissing postbaseline values up to 30 days after last dosing date.

In addition to the summary above, the Graded laboratory abnormalities and Grade 3 or 4 laboratory abnormalities will also be summarized using only the data from GS-US-401-1787.

A by-subject listing of treatment-emergent Grade 3 or 4 laboratory abnormalities and marked laboratory abnormalities will be provided by subject ID number and visit in chronological order. This listing will include all test results that were collected throughout the study for the lab test of interest, with all applicable severity grades or abnormal flags displayed.

#### 7.2.3. Liver-related Laboratory Evaluations

Liver-related abnormalities after initial study drug dosing will be examined and summarized using the number and percentage of subjects who were reported to have the following laboratory test values for postbaseline measurements:

- Aspartate aminotransferase (AST): (a) > 3 times of the upper limit of reference range (ULN);
   (b) > 5 x ULN; (c) > 10 x ULN; (d) > 20 x ULN
- Alanine aminotransferase (ALT): (a) > 3 x ULN; (b) > 5 x ULN; (c) > 10 x ULN;
   (d) > 20 x ULN
- AST or ALT: (a)  $> 3 \times \text{ULN}$ ; (b)  $> 5 \times \text{ULN}$ ; (c)  $> 10 \times \text{ULN}$ ; (d)  $> 20 \times \text{ULN}$
- Total bilirubin: > 2 x ULN
- Alkaline phosphatase (ALP) > 1.5 x ULN
- AST or ALT > 3 x ULN and total bilirubin: (a) > 1.5 x ULN; (b) > 2 x ULN

The summary will include data from all postbaseline visits up to 30 days after the last dose of study drug. For individual laboratory tests, subjects will be counted once based on the most severe postbaseline values. For both the composite endpoint of AST or ALT and total bilirubin, subjects will be counted once when the criteria are met at the same postbaseline visit date. The denominator is the number of subjects in the Safety Analysis Set who have nonmissing postbaseline values of all relevant tests at the same postbaseline visit date. A listing of subjects who met at least 1 of the above criteria will be provided.

#### 7.2.4. Shifts Relative to the Baseline Value

Shift tables will be presented by showing change in severity grade from baseline to the worst postbaseline grade.

### 7.3. Body Weight and Vital Signs

Descriptive statistics will be provided by treatment group for body weight, BMI, and vital signs as follows:

- Baseline value
- Postbaseline maximum
- Postbaseline minimum
- Change and percent change from baseline to postbaseline maximum
- Change and percent change from baseline to postbaseline minimum

A baseline value will be defined as the last available value collected on or prior to the date/time of first dose of study drug in the parent study. Change from baseline to a postbaseline visit will be defined as the postbaseline value minus the baseline value. Body weight and vital signs measured at unscheduled visits will be included for the baseline value selection, and postbaseline maximum and minimum value selection.

A by-subject listing of vital signs will be provided by subject ID number and time point in chronological order. Body weight and BMI will be included in the vital signs listing, if space permits. If not, they will be provided separately.

#### 7.4. Prior and Concomitant Medications

Medications collected in the GS-US-401-1787 study will be coded using the current version of the World Health Organization (WHO) Drug dictionary. The coding of Medications collected in the parent study ONO-4059POE001 will be upversioned to the current version of WHODrug, and integrated with GS-US-401-1787 for analysis.

### 7.4.1. Prior Medications

Prior medications are defined as any medication taken before a subject took the first study drug of parent study.

Prior medications will be summarized by Anatomical Therapeutic Chemical (ATC) drug class Level 2 and preferred name using the number and percentage of subjects for each treatment group and overall. A subject reporting the same medication more than once will be counted only once when calculating the number and percentage of subjects who received that medication. The summary will be ordered alphabetically by ATC medical class and then by preferred term in order of descending overall frequency within each ATC medical class. For drugs with the same frequency, sorting will be done alphabetically.

For the purposes of analysis, any medication with a start date prior to the first dosing date of study drug will be included in the prior medication summary regardless of when the stop date is. If a partial start date is entered the medication will be considered prior unless the month and year (if day is missing) or year (if day and month are missing) of the start date are after the first dosing date. Medications with a completely missing start date will be included in the prior medication summary, unless otherwise specified.

Summaries will be based on the Safety Analysis Set. No formal statistical testing is planned.

#### 7.4.2. Concomitant Medications

Concomitant medications are defined as medications taken while a subject took study drug. Use of concomitant medications will be summarized by Anatomical Therapeutic Chemical (ATC) drug class Level 2 and preferred name using the number and percentage of subjects for each treatment group. A subject reporting the same medication more than once will be counted only once when calculating the number and percentage of subjects who received that medication. The summary will be ordered alphabetically by ATC medical class and then by preferred term in descending overall frequency within each ATC medical class. For drugs with the same frequency, sorting will be done alphabetically.

For the purposes of analysis, any medication with a start date prior to or on the first dosing date of study drug and continued to take after the first dosing date, or started after the first dosing date but prior to or on the last dosing date of study drug will be considered concomitant medications. Medications started and stopped on the same day as the first dosing date or the last dosing date of study drug will also be considered concomitant. Medications with a stop date prior to the date of first dosing date of study drug or a start date after the last dosing date of study drug will be excluded from the concomitant medication summary. If a partial stop date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) prior to the date of first study drug administration will be excluded from the concomitant medication summary. If a partial start date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) after the study drug stop date will be excluded from the concomitant medication summary. Medications with completely missing start and stop dates will be included in the concomitant medication summary, unless otherwise specified. Summaries will be based on the Safety Analysis Set. No formal statistical testing is planned.

All prior and concomitant medications (other than per-protocol study drugs) will be provided in a by-subject listing sorted by subject ID number and administration date in chronological order.

# 7.5. Electrocardiogram Results

Electrocardiogram (ECG) analysis results are intended to identify meaningful changes in the QT interval. If potential abnormalities of interest are identified, further analyses may be conducted.

A shift table of the investigators' assessment of ECG results at each visit compared with baseline values will be presented by treatment group using the following categories: normal; abnormal, not clinically significant; abnormal, clinically significant; or missing. The number and percentage of subjects in each cross-classification group of the shift table will be presented. Subjects with a missing value at baseline or postbaseline will not be included in the denominator for percentage calculation. No formal statistical testing is planned.

A by-subject listing for ECG assessment results will be provided by subject ID number and time point in chronological order.

### 7.6. Other Safety Measures

No additional safety measures are specified in the protocol.

# 7.7. Changes From Protocol-Specified Safety Analyses

There are no deviations from the protocol-specified safety analyses.

#### 8. PHARMACOKINETIC ANALYSES

### 8.1. Pharmacokinetics (PK) Sample Collection

Plasma samples for PK will be collected to measure concentrations of tirabrutinib at pre-dose of GS-US-401-1787 Cycles 2 and 3 only.

### 8.2. Statistical Analysis Methods

#### 8.2.1. Tirabrutinib Plasma Concentration

PK concentration data from GS-US-401-1787 will be summarized. PK analysis set will be grouped as specified in Section 3.2.

Tirabrutinib plasma concentration data will be summarized using descriptive statistics for subjects in the PK Analysis Set by time point and visit. Subjects in different dose levels will be presented separately. The sample size for each time point will be based on the number of subjects with nonmissing concentration data at that time point. The number of subjects with concentration BLQ will be presented for each time point. For summary statistics, BLQ values will be treated as 0 at predose and one-half of the lower limit of quantitation (LLOQ) for postdose time points.

The following table will be provided by disease type and dose level:

• Individual subject concentration data and summary statistics

Tirabrutinib plasma concentration data and PK sampling details will be listed for all subjects in the PK Analysis Set.

### 8.3. Changes From Protocol-Specified PK Analyses

There are no deviations from the protocol-specified pharmacokinetic analyses.

### 9. REFERENCES

- Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, et al. Revised response criteria for malignant lymphoma. J Clin Oncol 2007;25 (5):579-86.
- Hallek M, Cheson BD, Catovsky D, Caligaris-Cappio F, Dighiero G, Dohner H, et al. Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia: a report from the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) updating the National Cancer Institute-Working Group (NCI-WG) 1996 guidelines. Blood 2008;111 (12):5446-56.
- Owen RG, Kyle RA, Stone MJ, Rawstron AC, Leblond V, Merlini G, et al. Response assessment in Waldenstrom macroglobulinaemia: update from the VIth International Workshop. Br J Haematol 2013;160 (2):171-6.

# 10. SOFTWARE

SAS® Software Version 9.4. SAS Institute Inc., Cary, NC, USA.

# 11. SAP REVISION

| Revision Date<br>(DD MMM YYYY) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|
| 10 Apr 2020, version 2.0 | 1.2.2 | Update the 401-1787 study design to maximum duration of 5 years treatment, per the protocol amendment 5 dated 29 October 2019 | Align with protocol amendment 5 dated 29 October 2019 |
| 10 Apr 2020, version 2.0 | 2.1,<br>3.1.2,<br>6 | Administrative changes | Language clarification |
| 10 Apr 2020, version 2.0 | 6.2.2 | Added PFS follow-up time analysis | To add additional analysis per new Gilead oncology standard |
| 10 Apr 2020, version 2.0 | 6.2.2 | Revised the data imputation rule for incomplete date of anti-cancer therapy | Update per Gilead oncology standard |
| 10 Apr 2020, version 2.0 | 6.2.4 | Added OS follow-up time analysis | To add additional analysis per new Gilead oncology standard |
| 10 February 2021, version 3.0 | 4.4 | Added the section to provide how to handle special situations due to COVID-19 in the analysis | To assess the COVID-19 impact |
# 12. APPENDICES

| COVID-19 SMQ with Broad Scope |
|--------------------------------------------------------|
| Determining Missing and Virtual Visits Due to COVID-19 |
| Bleeding/Haemorrhage Medical Search Term |
| Hypersensitivity Medical Search Term |
| Cytopenia Medical Search Term |
| Cardiac arrhythmia Medical Search Term |
| Rash Medical Search Term |
| List of Laboratory Tests for Safety Summary |

## Appendix 1. COVID-19 SMQ with Broad Scope


#### **Appendix 2.** Determining Missing and Virtual Visits Due to COVID-19

This appendix describes the clinical trial site collection of COVID-19 data pertaining to missed/virtual visits and the data processing algorithm used to determine which visits were missing and which visits were virtual.

#### Data collection

A COVID-19 supplement to the eCRF Completion Guidelines (CCG) was provided by data management to instruct clinical trial sites with respect to data entry expectations pertaining to scenarios related to the COVID-19 pandemic. If a visit was missed, sites should enter "Visit missed due to COVID-19." If an in-person visit was conducted virtually, sites should enter "Virtual visit due to COVID-19."

#### Determination of Missed and Virtual visits

NLP was used to search the CRF comment fields to identify instances of "COVID-19" (or synonyms, see the table below) and "Virtual" (or synonyms, see the table below). The search terms are maintained in a global lookup table and can be modified to tune the NLP model. For any comments with COVID-19 search terms, assign "Missed visit" or "Virtual visit as follows:

- i. If COVID-19 terms are identified through NLP and the visit date is missing, then result is "Missed Visit"
- ii. If COVID-19 and Virtual terms are identified through NLP for a visit, then result is "Virtual Visit". When there are multiple records for the same subject and the same visit, NLP will be based on multiple records to ensure 1 unique category per subject per visit
- iii. Otherwise result is missing

# Examples of Search Terms for "COVID-19" and "Virtual" Used to Identify Missed and Virtual Visits

| Search Terms for "COVID-19" | Search Terms for "Virtual" |
|-----------------------------|----------------------------|
| COVID19 | VIRTUAL |
| CORONA | TELEMED |
| CORONAVIRUS | TELEHEALTH |
| PANDEMIC | TELEPHONE |
| OUTBREAK | REMOTE |
| CRISIS | TELEMEDICINE |
| LOCKDOWN | TELECONSULTATION |
| QUARANTINE | TELEPHONICALLY |
| SHELTER | PHONE |
| | HOME VISIT |
| | ZOOM |
| | SKYPE |

## Appendix 3. Bleeding/Haemorrhage Medical Search Term


#### Appendix 4. Hypersensitivity Medical Search Term


## **Appendix 5.** Cytopenia Medical Search Term


#### **Appendix 6.** Cardiac arrhythmia Medical Search Term


## Appendix 7. Rash Medical Search Term


## **Appendix 8.** List of Laboratory Tests for Safety Summary

| Serum Chemistry | Hematology |
|----------------------|-----------------|
| Albumin | WBC |
| Alkaline phosphatase | Hemoglobin |
| ALT | Hematocrit |
| Amylase | Platelet Count |
| AST | Basophils |
| Bicarbonate | Monocytes |
| BUN | Eosinophils |
| Calcium | Neutrophils |
| Chloride | Lymphocytes |
| Creatininea | Red Blood Cells |
| GGT | |
| Glucose <sup>b</sup> | |
| LDH | |
| Lipase | |
| Potassium | |
| Sodium | |
| Total bilirubin | |
| Total Protein | |
| Uric Acid | |

a Both creatinine and creatinine clearance rate will be included in the safety summary. Estimated creatinine clearance rate will be calculated based on the Cockcroft-Gault formula

b If fasting status is not unknown, non-fasting criteria will be applied for toxicity grading.

# SAP GS-US-401-1787 v3.0

# **ELECTRONIC SIGNATURES**

| Signed by | Meaning of Signature | Server Date<br>(dd-MMM-<br>yyyy hh:mm:ss) |
|---|---|---|
| PPD | Clinical Pharmacology<br>eSigned | 02-Mar-2021<br>19:51:40 |
| PPD | Clinical Research eSigned | 04-Mar-2021<br>01:56:25 |
| PPD | Biostatistics eSigned | 05-Mar-2021<br>07:32:28 |